CLINICAL TRIAL: NCT04319991
Title: The Clinical Evaluation of Probiotics Product in Patients With Various Functional Bowel Disorders and Helicobacter Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fooyin University (Other)
Responsible Party: Principal Investigator, Ching-Chiang, Lin, professor, Fooyin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FYH-IRB-108-07-01
Record Dates: First submitted 2020-03-06; First posted 2020-03-24 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Bowel Dysfunction; Helicobacter Pylori Infection
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Probiotics product
- Probiotics product (Experimental)
  Interventions: Dietary Supplement: Probiotics product

INTERVENTIONS:
Dietary Supplement: Probiotics product — This Probiotics product is a supplement containing several types of probiotics and prebiotics which has been marketed for years in Taiwan. Each sachet contains 3 grams granule. Take 1 sticks 3 times per day with or without water before meals.

SUMMARY:
People nowadays tend to have irregular diet and routine due to the stress at work. This condition may cause intestinal microflora imbalance, and in the long term may lead to constipation, diarrhea, gastroenteritis, gastric ulcer and other gastrointestinal diseases. Helicobacter pylori infection, which can trigger gastrointestinal inflammation and ulcer, is commonly treated by antibiotics. This treatment, however, can reduce the diversity of the intestinal microflora, causing diarrhea, flatulence and nausea. Clinical trials showed that probiotics and prebiotics supplementation could regulate gastrointestinal function, including alleviating constipation, ameliorating antibiotic-associated diarrhea and flatulence, enhancing the effect of H. pylori treatment, and restoring the balance of intestinal microflora. This Probiotics product is a supplement containing several types of probiotics and prebiotics which has been marketed for years. This project aims to observe the effectiveness of Probiotics product consumption by H. pylori-infected patients in relieving the gastrointestinal symptoms and restoring their intestinal microflora.

ELIGIBILITY:
Inclusion Criteria (PART I : For patients with bowel disorders):

* Constipation : Must include 2 or more of the following:

  * straining during at least 25% of defecations
  * lumpy or hard stools in at least 25% of defecations
  * sensation of incomplete evacuation for at least 25% of defecations
  * sensation of anorectal obstruction/blockage for at least 25% of defecations
  * manual maneuvers to facilitate at least 25% of defecations
  * fewer than 3 defecations per week
* Diarrhea :

  * the passage of 3 or more loose or liquid stools per day and lasting more than 1 week, or more frequently than is normal for the individual.

Inclusion Criteria (PART II : For patients with Helicobacter pylori infection):

* Campylobacter-like organism test (CLO test) positive

Exclusion Criteria (PART I & II)

* prior upper digestive tract surgery
* a history of cancer
* lactose intolerance
* allergy to penicillin
* prior antibiotics therapy in the last month
* prior probiotics supplement more than once a week in the last three weeks

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
The degree of microbiota correction or improvement by specific probiotic strain(s) | Changes from Baseline Fecal Microbiota at 4 weeks
  16S ribosomal RNA (rRNA) sequencing is a common amplicon sequencing methods used to identify and compare bacteria present within a given sample. 16S rRNA gene sequencing is a well-established method for comparing sample phylogeny and taxonomy from complex microbiomes.
Questionnaire to assess the severity and frequency of symptoms was reported | Changes from Baseline GSRS at 4 weeks
  The Gastrointestinal Symptom Rating Scale (GSRS) is a disease-specific questionnaire of 15 items to assess the severity and frequency of symptoms was reported; GSRS uses a 7-point Likert scale ranging from 1 = no problem to 7 = a very severe problem.

CONTACTS AND LOCATIONS:
Locations (1):
- Fooyin University Hospital, Pingtung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided